CLINICAL TRIAL: NCT01533194
Title: A Phase 1 Study of Reolysin Alone in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Viral Therapy in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-00248; NCI-2012-00248 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000724857; 2011C0141; 9030; OSU 11148 (Other: Ohio State University Comprehensive Cancer Center); 9030 (Other: CTEP); P30CA016058 (NIH); U01CA076576 (NIH)
Record Dates: First submitted 2012-02-11; First posted 2012-02-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2014-12

CONDITIONS: Light Chain Deposition Disease; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — reolysin

ARMS (1):
- Treatment (wild-type reovirus) (Experimental): Patients receive wild-type reovirus IV over 60 minutes on days 1-5. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Diagnostic Laboratory Biomarker Analysis; Biological: Wild-type Reovirus

INTERVENTIONS:
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Biological: Wild-type Reovirus — Given IV
  Other Names: Reolysin

SUMMARY:
This pilot phase I trial studies the side effects and the best dose of giving viral therapy to patients with relapsed or refractory multiple myeloma. Viral therapy, such as wild-type reovirus, may be able to kill cancer cells without damaging normal cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine safety and tolerability of Reolysin in patients with relapsed multiple myeloma.

II. Obtain evidence of Reovirus replication by immunohistochemical co-localization of Reovirus and tubulin staining in marrow clot sections obtained on cycle 1 day 8.

SECONDARY OBJECTIVES:

I. Obtain preliminary data on response as determined by International Myeloma Working Group criteria after infusion of Reolysin as a single agent. (Clinical) II. Obtain pilot overall and progression free survival data for all treated patients. (Clinical) III. Assess neutralizing anti-reovirus assay (NARA) results on days 1, 8, 15, and once days 22-28 during cycle 1. (Correlative) IV. Assess feasibility of staining for RAF/MEK/ERK in CD138+ cells using marrow clot sections obtained from pre-treatment specimen. (Correlative) V. Cryopreserve PBMCs for future ancillary studies focused initially on lymphocyte subset(s) and myeloid derived suppressor cell changes after Reolysin infusion during cycle 1. (Correlative) VI. Cryopreserve CD138+-selected cells at screening and after treatment for future ancillary studies of genetic and epigenetic changes focused in part on endoplasmic reticulum (ER) stress. (Correlative)

OUTLINE: This is a dose-escalation study.

Patients receive wild-type reovirus IV over 60 minutes on days 1-5. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo bone marrow aspirate at baseline and periodically during study for RAF/MEK/ERK expression and wild-type reovirus replication analysis by immunohistochemistry. Blood and cryopreserved CD138+ selected cell samples are also collected for future ancillary studies.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have relapsed or refractory myeloma that fits or did fit IMWG diagnostic criteria for symptomatic myeloma (although new or worsening end-organ damage is not required to be eligible) as defined below:

  * Presence of ≥ 10% clonal bone marrow plasma cells
  * Presence of serum and/or urinary measurable monoclonal protein or light chains
  * Evidence of any end-organ damage criteria listed below [at any time] attributed to the patient's myeloma:

    * Hypercalcemia: Serum calcium > 11.5 mg/dL
    * Renal insufficiency: Serum creatinine > 2 mg/dL
    * Anemia > 2 g/dL below the lower limit of normal or a hemoglobin value < 10 g/dL
    * Bone lesions: Lytic lesions, severe osteopenia, or pathologic fractures
* Subject must have measurable disease defined as any of the following:

  * Serum monoclonal protein > 500 mg/dL by protein electrophoresis
  * > 200 mg of monoclonal protein in the urine on 24-hour electrophoresis
  * Serum immunoglobulin free light chain ≥ 100 mg/L AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
* Patients must have received at least one prior antineoplastic therapy and must have progressed
* No standard therapy is available or patient declines such options
* Prior autologous and/or allogeneic transplant is permitted although transplant must have occurred greater than 90 days prior to registration
* Adverse events from prior therapy must have recovered to no greater than grade 1 with the exception of grade 2 neuropathy
* Prior radiation is permitted; however, at least 4 weeks must have elapsed since the completion of prior radiation therapy and patients must have recovered from all radiation-associated toxicities to no greater than grade 1 at the time of registration
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%); patients with lower performance status based solely on bone pain secondary to multiple myeloma will be eligible
* Life expectancy of greater than 3 months
* Absolute neutrophil count (ANC) ≥ 1,000/μL
* Platelet count ≥ 50,000/μL
* Hemoglobin > 8 g/dL
* Total bilirubin < 1.5 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 times the institutional upper limit of normal.
* Able to understand and willing to sign a written informed consent document
* Patients must be able to avoid direct contact with pregnant or nursing women, infants, and immunocompromised individuals during the five days of Reolysin treatment and for two days after
* Patients must not have known immunodeficiency virus (HIV) infection or active hepatitis B or C infections
* For patients with a history of congestive heart failure, systolic cardiac function must be assessed at screening and left ventricular ejection fraction (LVEF) ≥ 50%
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL prior to starting therapy and prior to beginning another course (if applicable)
* FCBP and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* The patient must be willing to comply with fertility requirements as below:

  * Male patients must agree to use an adequate method of contraception for the duration of the study and for 90 days afterwards
  * Female patients must be either postmenopausal, free from menses ≥ 2 years, surgically sterilized, willing to use two adequate barrier methods of contraception to prevent pregnancy, or agree to abstain from heterosexual activity starting with screening and for 90 days afterwards
  * Patients must agree not to donate blood or sperm/ova during the course of taking protocol therapy and for at least 4 weeks after stopping treatment
* No patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study

  * Patients may be receiving concomitant therapy with bisphosphonates and low-dose corticosteroids (e.g., prednisone up to but no more than 10 mg by mouth daily or its equivalent) for symptom management and comorbid conditions; doses of corticosteroid should be stable for at least 7 days prior to study treatment
* No patients who are receiving any other investigational agents
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, myocardial infarction in the preceding 6 months, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study
* No patients with a "currently active" second malignancy that, in the opinion of the principal investigator, will interfere with patient participation, increase patient risk, shorten survival to < 1 year, or confound data interpretation
* No POEMS syndrome
* No concurrent use of complementary or alternative medicines that, in the opinion of the principal investigator, would confound the interpretation of toxicities and/or antitumor activity of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Associated adverse events based on Common Terminology Criteria for Adverse Events (CTCAE) criteria and tolerability of wild-type reovirus | Up to 4 weeks post-treatment
  The number and severity of toxicity incidents will indicate the level of tolerance for Reolysin in the treatment of relapsed/refractory multiple myeloma. Toxicities will be evaluated using the CTCAE v. 4 standard toxicity grading. Frequency distributions and other descriptive measures will form the basis of the analysis of these variables.
Maximum-tolerated dose level | 28 days
  The number and severity of toxicity incidents will indicate the level of tolerance for Reolysin in the treatment of relapsed/refractory multiple myeloma. Toxicities will be evaluated using the CTCAE v. 4 standard toxicity grading. Frequency distributions and other descriptive measures will form the basis of the analysis of these variables.

SECONDARY OUTCOMES:
Duration of response | Up to 2 years
  Defined as the duration from first observation of partial response to the time of disease progression (taking as a reference for progressive disease the smallest measurements recorded since treatment started), with deaths due to other causes other than progression censored. This includes only patients with confirmed responses, and the date at which the response status was first observed rather than the date of confirmation is used as the start date.
Objective response rate | Up to 4 weeks post-treatment
  Will evaluate clinical benefit endpoint described as that portion of patients experiencing CR, VGPR, or PR. The objective response rate will be analyzed by using a 95% confidence interval for the proportion responding at trial closure in the treated population.
Progression-free survival | From start of treatment to disease progression or death, regardless of cause of death, whichever comes first, assessed up to 2 years
Time to progression | Time from the start of the treatment until the criteria for disease progression are met, assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hofmeister, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States